CLINICAL TRIAL: NCT04426721
Title: Intra-articular Oxygen-ozone Therapy for the Treatment of Knee Osteoarthritis: a Randomized, Double-blind, Clinical Trial Compared With Hyaluronic Acid
Brief Title: Intra-articular Oxygen-ozone Therapy for the Treatment of Knee Osteoarthritis Compared With Hyaluronic Acid
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Humanitas Clinical and Research Center (Other)
Responsible Party: Principal Investigator, Cristiano Sconza, Principal Investigator, Humanitas Clinical and Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OZKOA1
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Knee Osteoarthritis
Keywords: Oxygene-Ozone; Ozone; Hyaluronic acid; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Ozone; Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ozone (Experimental): Participant will receive an intraarticular injection of oxygen-ozone, once a week for three weeks. During procedure a clear ultrasound image is to be taken to document needle placement in the synovial space. The injector may choose the position of the knee (e.g., extended or bent) and the approach for the injection (e.g., medial or lateral).
  Interventions: Drug: Ozone
- Hyaluronic acid (Active Comparator): Participant will receive an intraarticular injection of hyaluronic acid, once a week for three weeks. During procedure a clear ultrasound image is to be taken to document needle placement in the synovial space. The injector may choose the position of the knee (e.g., extended or bent) and the approach for the injection (e.g., medial or lateral).
  Interventions: Drug: Hyaluronic Acid

INTERVENTIONS:
Drug: Ozone — 10 cc of oxygen-ozone
  Other Names: Oxygene-Ozone therapy; O2-O3
  Arms: Ozone
Drug: Hyaluronic Acid — Sinovial forte 32 mg\2ml
  Other Names: Sinovial forte
  Arms: Hyaluronic acid

SUMMARY:
Knee osteoarthritis is a very common pathology, characterized by pain, stiffness and functional deficit. The various therapeutic options used include anti-inflammatory drug treatment, physiokinesitherapy, minimally invasive procedures and, finally, in non-responsive cases, surgical treatment. To date, several studies have been conducted on the intra-articular use of oxygen-ozone in knee osteoarthritis and its potential therapeutic benefits. However, the methodological quality of the RCTs available in the literature is not satisfactory, so it is necessary to define a standardized protocol for therapy and procedures. The aim of this study will be to develop a rigorous protocol to evaluate the effectiveness of intra-articular oxygen-ozone therapy (OOT) in knee osteoarthritis and compare it with injection therapy with hyaluronic acid (HA), currently widely used in the treatment of knee osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis is a degenerative condition that causes pain, impaired function and affects daily activities. In knee osteoarthritis, there is destruction of cartilage and subchondral bone, with the consequent narrowing of articular space. Besides the biomechanical factors, trauma and obesity; it is believed that inflammation plays an important role. Treatment options for painful knee osteoarthritis are often unsatisfactory, as represented by 40% of patients reporting persisting postoperative pain following total knee arthroplasty . There are no currently approved knee osteoarthritis treatments capable of slowing OA-related structural progression, so the main goals of the conservative treatment are to provide symptomatic relief, improve joint function, and delay surgical intervention. One of the main actions of intra-articular treatments, ranging from corticosteroids to hyaluronic acid (HA) and biologic products is to reduce inflammatory distress within the joint. In recent years, there has been a growing interest in the effects of ozone, which can be safely delivered intra-articularly and whose use is in constant increase in an outpatient setting due to the ease of preparation methods. From the literature, it is widely accepted that ozone has the biological properties of inducing analgesia, anti-inflammatory, and antioxidant effects mediated by activating the cellular metabolism and inhibiting prostaglandin synthesis, reduce edema and inflammation, and therefore reduce pain and improves function in knee osteoarthritis. Intra-articular oxygen-ozone has been used in the medical domain for several decades. Although some articles have reported promising results on the effectiveness of oxygen-ozone in knee osteoarthritis, the evidence is however low . Currently, few RCTs have compared the efficacy and safety of ozone therapy versus HA intra-articular injections in patients affected by knee osteoarthritis. This study will compare the efficacy of OOT injection to HA in patients with symptomatic OA in one knee, who have failed at least one prior conservative OA therapy (e.g. physiotherapy, simple analgesics). This will be done using a double blind, randomized controlled trial with study subjects receiving a cycle of three injection of OOT or HA. The primary efficacy measure will be pain measured by the WOMAC LK 3.1 scale; other measures of efficacy will include function, stiffness, and quality of life. In addition to clinical efficacy measures, safety will be assessed by tracking adverse events. During screening, potential subjects who provide informed consent will be assessed for eligibility. Screening will consist in checking the presence of inclusion and exclusion criteria, including a WOMAC LK 3.1 pain subscale score ≥ 9 and ≤ 19 and by providing objective physiological evidence of OA using the Kellgren-Lawrence scale (assessed from radiographs). Subjects will also provide demographic and medication use information. Baseline X-ray and MRI will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 18 years of age at time of screening.
2. Ability to comply with study procedures and visit schedules and able to follow oral and written instructions.
3. Patients with symptomatic OA in one knee from 3 months
4. A standing knee radiograph showing a K-L grade of 2 to 3 and an absence of severe osteoarthritis (defined as advanced stage osteoarthritis, including large osteophytes, chronic fractures or bone remodeling, severe deformity or bone attrition, and/or bone-on-bone contact indicative of severe osteoarthritis/full thickness cartilage loss).
5. Body mass index ≤ 40 kg/m2.
6. A WOMAC LK 3.1 pain subscale total score ≥ 9 and ≤ 19.
7. Has undergone at least one prior conservative OA treatment (e.g. physical therapy, simple analgesics).
8. Signed an ethics committee-reviewed an approved informed consent form.

Exclusion Criteria:

1. Presence of clinically observed active infection or severe inflammation in the index knee joint or skin disease/breakdown or infection in the area of the planned injection site of the index knee.
2. Presence of symptomatic OA in the non-study knee at screening; if unclear then the WOMAC LK 3.1 pain subscale for the non-index knee must be ≤ 5.0.
3. Diagnosed with rheumatoid arthritis, Reiter's syndrome, psoriatic arthritis, gout, ankylosing spondylitis, or arthritis secondary to other inflammatory diseases; Human Immunodeficiency Virus (HIV), viral hepatitis; chondrocalcinosis, Paget's disease, or villonodular synovitis.
4. Diagnosed with leukemia, known presence of metastatic malignant cells, or ongoing or planned chemotherapeutic treatment.
5. Disease of spine, hip or other lower extremity joints judged by the investigator to be contributing to the pain in the index knee (e.g. sciatica, nerve pain, hip OA). Note: Patients with contralateral knee replacement, or hip replacement in either hip, may be enrolled provided there is sufficient pain relief after knee replacement or hip replacement that analgesics are not required.
6. Untreated symptomatic injury of the index knee (e.g., acute traumatic injury, anterior cruciate ligament injury, clinically symptomatic meniscus injury characterized by mechanical issue such as locking or catching).
7. Presence of surgical hardware or other foreign body intended to treat arthritis or cartilage-related pathology in the index knee. Note: this does not include small hardware (e.g. screws).
8. Presence of venous or lymphatic stasis in the index leg.
9. Orally administered systemic steroid use within 2 weeks prior to screening
10. Planned/anticipated surgery of the index knee during the study period.
11. Major surgery of the index knee within 12 months prior to screening.
12. Minor surgery (e.g. arthroscopy) of the index knee within 6 months prior to screening.
13. Any documented clinically significant degree of cognitive impairment or other condition, finding, or psychiatric illness at screening, which, in the opinion of the investigator, could compromise patient safety or interfere with the assessment of the safety and treatment effects of the study injection.
14. Pregnant or nursing mothers or women planning to become pregnant during the time they will be participating in the study.
15. Know hypersensitivity (allergy) to hyaluronan (sodium hyaluronate) preparations.
16. Previously documented failed treatment with OOT or Sinovial
17. Known drug or alcohol dependence currently or within the last year.
18. Use of any investigational drug or device within 30 days prior to screening.
19. Use of any investigational biologics within 60 days prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index using the Likert scale, Version 3.1, Pain subscale (WOMAC LK 3.1) | 3 months
  Assessment of pain. Score range 0-20. Higher scores indicate worse pain.

SECONDARY OUTCOMES:
The Western Ontario and McMaster Universities Osteoarthritis Index using the Likert scale, Version 3.1(WOMAC LK 3.1) | 1,3,6,12 months
  Assessment of pain, stiffness and function. Score range 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Higher scores indicate worse pain, stiffness, and functional limitations.
Numeric Rating Scale (NRS) | 1,3,6,12 months
  Assessment of pain. Score range 0-10. Higher scores indicate worse pain.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 1,3,6,12 months
  Assessment of Pain, other Symptoms, Function in daily living, Function in Sport and Recreation, and knee-related Quality of Life (QOL). Score range 0-100, with zero representing extreme knee problems and 100 representing no knee problems

CONTACTS AND LOCATIONS:
Overall Officials: Cristiano Sconza, MD, Principal Investigator — Humanitas Clinical and Research Hospital; Berardo Di Matteo, MD, PhD, Study Chair — Humanitas Clinical and Research Hospital
Locations (1):
- Humanitas Clinical and Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided